CLINICAL TRIAL: NCT07123623
Title: The Effect of Couples' Participation in Childbirth Preparation Education on Pregnant Women's Perceived Spousal Support, Fear of Childbirth, and Self-Efficacy
Status: Recruiting | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Other Study IDs: Atlas Universty
Record Dates: First submitted 2025-04-09; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: The Effect of Couples' Participation in Childbirth Preparation Education on Pregnant Women's Perceived Spousal Support, Fear of Childbirth, and Self-Efficacy
Keywords: Childbirth Preparation Training, Father Involvement, Fear of Childbirth, Partner Support, Childbirth Self-Efficacy.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mothers who have not received prenatal education
- Expectant mothers undergoing childbirth preparation training
- Expectant parents undergoing childbirth preparation training

SUMMARY:
Fear of childbirth can be defined as approaching the process of giving birth with fear and anxiety. The aim of prenatal education is to help expectant mothers develop positive feelings towards childbirth and to foster a sense of security.

ELIGIBILITY:
Inclusion Criteria:

* Having applied to the specified institution within the study period
* Willingness to participate in the study
* Having at least a primary school education
* Pregnant women over the age of 18
* Being over the 20th week of pregnancy
* Having given birth vaginally at least once (for the multiparous group)
* Having a singleton pregnancy

Exclusion Criteria:

* Those who do not consent to participate in the study
* Pregnant women with a gestational age of less than 20 weeks
* Individuals with communication impairments
* Individuals with sensory-perceptual disorders
* Individuals with any psychiatric illness
* Pregnant women under the age of 18
* Pregnant women who have not completed at least primary school education.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: Expectant mothers over the age of 18 who have completed their 20th week of pregnancy and have applied to the hospital where the study will be conducted.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Spousal Support Scale(SSS), | A training program consisting of 4 weeks
  The aim of this study is to determine the effect of couples' participation in childbirth preparation education on pregnant women's perceived spousal support, fear of childbirth, and self-efficacy. Based on the scales used, it is expected that as pregnant women's fear of childbirth decreases, their perceived spousal support will increase.
  H2: Couples' participation in childbirth preparation education has an effect on perceived spousal support.
  The Spousal Support Scale (SSS), developed to assess the level of support between partners, consists of a total of 27 items. The scale is a 3-point Likert-type measurement tool, with items scored as "true for me" = 3, "partly true" = 2, and "not true for me" = 1. Items 10, 20, and 24 are reverse scored. The total score that can be obtained from the scale ranges between 27 and 81, with higher scores indicating higher levels of spousal support.
Wijma Delivery Expectancy/Experience Questionnaire Version A | A training program consisting of 4 weeks
  The aim of this study is to determine the effect of couples' participation in childbirth preparation classes on pregnant women's fear of childbirth, perceived spousal support, and childbirth self-efficacy. According to the scales used, it is expected that as pregnant women's fear of childbirth decreases, their perceived spousal support and childbirth self-efficacy will increase.
  H1: Couples' participation in childbirth preparation classes together with pregnant women has an effect on the pregnant women's fear of childbirth.
  The Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) is a 33-item scale. Responses are rated on a 6-point Likert scale ranging from 0 to 5, where 0 means "completely" and 5 means "not at all." The minimum possible score on the scale is 0 and the maximum is 165, with higher total scores indicating higher levels of fear. The W-DEQ is used to obtain a fear score related to childbirth.
Birth Self-Efficacy Scale Short Form (BSES-SF32) | A training program consisting of 4 weeks
  The aim of this study is to determine the effect of couples' participation in childbirth preparation education on pregnant women's perceived spousal support, fear of childbirth, and self-efficacy. Based on the scales used, it is expected that as pregnant women's fear of childbirth decreases, their childbirth self-efficacy will increase.
  H3: Couples' participation in childbirth preparation classes has an effect on pregnant women's childbirth self-efficacy.
  The scale was developed to measure women's self-efficacy regarding the childbirth process. It consists of 32 items and two sub-dimensions: efficacy expectancy and outcome expectancy. Scores from the subscales range between 16 and 160. Higher scores on the subscales indicate higher efficacy and outcome expectancy related to childbirth. The Cronbach's alpha coefficient of the scale is 0.90.
Spousal Support Scale(SSS), The Wijma Delivery Expectancy/Experience Questionnaire Version A (W-DEQ), Birth Self-Efficacy Scale Short Form (BSES-SF32) | A training program consisting of 4 weeks
  ChatGPT:
  The aim of this study is to determine the effect of couples' participation in childbirth preparation education on pregnant women's perceived spousal support, fear of childbirth, and childbirth self-efficacy. Based on the scales used, it is expected that as pregnant women's fear of childbirth decreases, their perceived spousal support and childbirth self-efficacy will increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas Universty, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aguilera-Martin A, Galvez-Lara M, Blanco-Ruiz M, Garcia-Torres F. Psychological, educational, and alternative interventions for reducing fear of childbirth in pregnant women: A systematic review. J Clin Psychol. 2021 Mar;77(3):525-555. doi: 10.1002/jclp.23071. Epub 2020 Oct 20. PMID 33078851
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30693793/https://www.turkailehekderg.org/jvi.aspx?un=TAHD-98608&volume=26&issue=1https://doi.org/10.1080/0167482X.2017.1398230https://dergipark.org.tr/tr/download/article-file/200064